CLINICAL TRIAL: NCT02478229
Title: Early Treatment With Sofosbuvir (SOF) and Ledipasvir (LDV) to Prevent HCV Recurrence After Liver Transplantation (OLT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty recruiting patients
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-8883-A
Record Dates: First submitted 2015-06-05; First posted 2015-06-23 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C Viral Infection
Keywords: Liver transplant; Genotype 1 HCV infection; Sofosbuvir (SOF)/ Ledipasvir (LDV); Sustained virological response (SVR12 )
MeSH Terms: interventions — Sofosbuvir; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOF and LDV (Experimental): Single arm: All participants will be started on Sofosbuvir (SOF) 400 mg and Ledipasvir (LDV) 90 mg as a fixed dose combination (FDC) tablet p.o. once daily with or without food starting at the time of liver transplantation (OLT), i.e. first doses given immediately prior to OLT, and continuing for 12 weeks.
  Interventions: Drug: Sofosbuvir (SOF) and Ledipasvir (LDV)

INTERVENTIONS:
Drug: Sofosbuvir (SOF) and Ledipasvir (LDV)

SUMMARY:
The study is a single centre, single arm, open-label, proof of concept study enrolling 20 adult primary liver transplant recipients with genotype 1 HCV infection. Subjects will receive Sofosbuvir (SOF) and Ledipasvir (LDV) starting at time of liver transplantation (OLT) and continues for 12 weeks. Subjects will be receive 24 week post-treatment follow up.

DETAILED DESCRIPTION:
Hepatitis C viral infection (HCV) leading to end-stage liver disease is the leading indication for liver transplant worldwide. HCV recurrence following liver transplantation is universal, associated with 100-fold increase in viremia levels, and runs at an accelerated course, leading to graft cirrhosis in up to 30% of patients within 5 years. Successful eradication of HCV post transplant normalizes the long term survival of HCV positive liver transplant recipients. This study aims to treat HCV infection starting at the time of transplant. The study is a single centre, single arm, open-label,proof of concept study enrolling 20 adult primary liver transplant recipients with genotype 1 HCV infection. Subjects will receive Sofosbuvir (SOF) 400 mg and Ledipasvir (LDV) 90 mg as a fixed dose combination (FDC) tablet starting at time of liver transplantation (OLT) and continues for 12 weeks. Subjects will receive 24 week post-treatment follow up. The study will investigate if the patient has achieved sustained virological response (SVR) 12 weeks after cessation of treatment (SVR12). Furthermore, safety and efficacy of this treatment regimen beginning at the time of transplant will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a first (primary) live or deceased (after brain or cardiac death) donor liver transplant
* Willing and able to provide written informed consent
* Male or Female, age 18-70 years old
* Medical MELD score ≤30 at time of transplant (calculated based on serum bilirubin, creatinine and INR, i.e. not taking exception points into account)
* Quantifiable HCV RNA at time of listing or transplant evaluation
* HCV genotype 1a or 1b infection
* Female patients must have a negative pregnancy test at enrolment

Exclusion Criteria:

* Liver re-transplantation
* Recipients of multiple solid organ transplants
* Estimated GFR <30ml/min at time of transplant
* Participants transplanted for fulminant hepatic failure
* Participants co-infected with HBV or HIV
* Previous treatment with a Sofosbuvir or Ledipasvir containing regimen
* Participation in an interventional clinical trial within 1 month prior to enrolment
* Known allergies or hypersensitivity to Sofosbuvir or Ledipasvir
* Pregnancy and/or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Sustained Virological Response (SVR12) | 12 weeks after cessation of treatment
  Defined as HCV RNA in serum below lower limit of quantification (LLOQ)

SECONDARY OUTCOMES:
Sustained Virological Response (SVR24) | 24 weeks after cessation of treatment
  Defined as HCV RNA in serum below lower limit of quantification (LLOQ)

OTHER OUTCOMES:
Virological Relapse | 12 weeks after cessation of treatment or 24 weeks after cessation of treatment (becoming quantifiable again at 12 (relapse 12) or 24 (relapse 24) weeks after cessation of treatment, respectively)
  Defined as HCV RNA in serum below lower limit of quantification (LLOQ)

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Renner, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Afdhal N, Reddy KR, Nelson DR, Lawitz E, Gordon SC, Schiff E, Nahass R, Ghalib R, Gitlin N, Herring R, Lalezari J, Younes ZH, Pockros PJ, Di Bisceglie AM, Arora S, Subramanian GM, Zhu Y, Dvory-Sobol H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Sulkowski M, Kwo P; ION-2 Investigators. Ledipasvir and sofosbuvir for previously treated HCV genotype 1 infection. N Engl J Med. 2014 Apr 17;370(16):1483-93. doi: 10.1056/NEJMoa1316366. Epub 2014 Apr 11. PMID 24725238
- [Background] Bzowej N, Nelson DR, Terrault NA, Everson GT, Teng LL, Prabhakar A, Charlton MR; PHOENIX Study Group. PHOENIX: A randomized controlled trial of peginterferon alfa-2a plus ribavirin as a prophylactic treatment after liver transplantation for hepatitis C virus. Liver Transpl. 2011 May;17(5):528-38. doi: 10.1002/lt.22271. PMID 21506241
- [Background] Gane EJ, Stedman CA, Hyland RH, Ding X, Svarovskaia E, Symonds WT, Hindes RG, Berrey MM. Nucleotide polymerase inhibitor sofosbuvir plus ribavirin for hepatitis C. N Engl J Med. 2013 Jan 3;368(1):34-44. doi: 10.1056/NEJMoa1208953. PMID 23281974
- [Background] Osinusi A, Meissner EG, Lee YJ, Bon D, Heytens L, Nelson A, Sneller M, Kohli A, Barrett L, Proschan M, Herrmann E, Shivakumar B, Gu W, Kwan R, Teferi G, Talwani R, Silk R, Kotb C, Wroblewski S, Fishbein D, Dewar R, Highbarger H, Zhang X, Kleiner D, Wood BJ, Chavez J, Symonds WT, Subramanian M, McHutchison J, Polis MA, Fauci AS, Masur H, Kottilil S. Sofosbuvir and ribavirin for hepatitis C genotype 1 in patients with unfavorable treatment characteristics: a randomized clinical trial. JAMA. 2013 Aug 28;310(8):804-11. doi: 10.1001/jama.2013.109309. PMID 23982366
- [Background] Selzner N, Renner EL, Selzner M, Adeyi O, Kashfi A, Therapondos G, Girgrah N, Herath C, Levy GA, Lilly L. Antiviral treatment of recurrent hepatitis C after liver transplantation: predictors of response and long-term outcome. Transplantation. 2009 Nov 27;88(10):1214-21. doi: 10.1097/TP.0b013e3181bd783c. PMID 19935376
- [Background] Sulkowski MS, Gardiner DF, Rodriguez-Torres M, Reddy KR, Hassanein T, Jacobson I, Lawitz E, Lok AS, Hinestrosa F, Thuluvath PJ, Schwartz H, Nelson DR, Everson GT, Eley T, Wind-Rotolo M, Huang SP, Gao M, Hernandez D, McPhee F, Sherman D, Hindes R, Symonds W, Pasquinelli C, Grasela DM; AI444040 Study Group. Daclatasvir plus sofosbuvir for previously treated or untreated chronic HCV infection. N Engl J Med. 2014 Jan 16;370(3):211-21. doi: 10.1056/NEJMoa1306218. PMID 24428467
- [Background] Tanaka T, Therapondos G, Selzner N, Renner EL, Lilly LB. Serum aspartate aminotransferase levels and previous histopathological findings enable reduction of protocol liver biopsies after liver transplantation for hepatitis C. Can J Gastroenterol. 2013 Mar;27(3):131-6. doi: 10.1155/2013/904636. PMID 23516677
- [Background] Tanaka T, Benmousa A, Marquez M, Therapondos G, Renner EL, Lilly LB. The long-term efficacy of nucleos(t)ide analog plus a year of low-dose HBIG to prevent HBV recurrence post-liver transplantation. Clin Transplant. 2012 Sep-Oct;26(5):E561-9. doi: 10.1111/ctr.12022. PMID 23061767